CLINICAL TRIAL: NCT02229630
Title: Prognostic Value of Diffusion-weighted Cerebral MRI in Prenatal Evaluation of Foetuses With Intra Uterine Growth Restriction.
Brief Title: Diffusion-weighted Cerebral MRI and Intra Uterine Growth Restriction.
Acronym: REDIFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P130915; IDRCB: 2014-A00640-47
Record Dates: First submitted 2014-07-17; First posted 2014-09-01 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pregnant Women With Foetuses Presenting With Intra-uterine Growth Restriction
Keywords: intra-uterine growth restriction; MRI; apparent diffusion coefficient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregnant women (Experimental): Foetuses with intra-uterine growth restriction, between 28 and 32 weeks of gestation, with an estimated foetal weight < 5th percentile (Hadlock calculator)
  Interventions: Radiation: Pregnant women with intra-uterine growth restricted Foetuses

INTERVENTIONS:
Radiation: Pregnant women with intra-uterine growth restricted Foetuses — Diffusion-weighted cerebral MRI before 32 weeks of gestation
  Other Names: cerebral MRI

SUMMARY:
The purpose of this study is to compare the apparent diffusion coefficient in the frontal lobe of foetuses with intra-uterine growth restriction and poor neonatal outcome compared with foetuses with intra-uterine growth restriction and a good neonatal outcome.

DETAILED DESCRIPTION:
Intra-uterine growth restriction is associated with an increased risk of perinatal morbimortality. The objective of foetal monitoring is to assess foetal growth, foetal well-being and to evaluate ability to adapt to chronic hypoxia.

The primary objective in antenatal care is to ischemic cerebral lesions. However, there is currently no relevant prenatal exam predictive for the risk of such lesions.

Foetal cerebral MRI could highlight changes in Apparent Diffusion Coefficient (ADC) in some frontal cerebral territories in foetuses with intra-uterine growth restriction and poor neonatal outcome.

These changes could be associated with a transient cerebral ischemia. The study of ADC could be a useful tool in the prognostic evaluation of these foetuses.

ELIGIBILITY:
Inclusion Criteria:

* single pregnancy
* estimated foetal weight ≤ 5th percentile
* agreeing to participate
* women age ≥ 18 years of age, speaking and understanding French language
* covered by the French social security system

Exclusion Criteria:

* foetal malformation or foetal karyotype abnormal
* infectious foetopathy
* multiple pregnancy
* refusal to participate
* pregnant women aged < 18 years old
* pregnant women not understanding or speaking French language
* not covered by French social security
* contraindication to MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2017-10-29 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Poor neonatal status | At birth
  Neonatal death; Apgar score < 7 at 5 min, immediate transfer to neonatal resuscitation unit; cordon arterial pH < 7.10

SECONDARY OUTCOMES:
Poor neonatal status | until 30 days of life
  Necrositing enterocolitis with need for surgical intervention; convulsions; intraventricular haemorrhage (type I to IV); periventricular leukomalacia (diagnosed by MRI); transfer to neonatal intensive care unit
Neonatal status at neonatology unit discharge | up to 20 weeks
  Neurological status: normal / abnormal; need in O2: Yes/No
Neurological development | At 2 years of age (adjusted age)
  Age and stages questionnaire (ASQ)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Jouannic, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Armand Trousseau, Paris, France

REFERENCES:
- [Background] Xu E, Jouannic JM, Alison M, Ancel PY, Friszer S, Rousseau J, Guilbaud L, Adamsbaum C, Goffinet F, Blondiaux E. Analysis of MRI brain biometrics in fetuses monitored for intra uterine growth restriction and their prognostic value: Results of a prospective multicenter study. Eur J Obstet Gynecol Reprod Biol. 2024 Jul;298:91-97. doi: 10.1016/j.ejogrb.2024.04.043. Epub 2024 Apr 30. PMID 38735121
- [Background] Jouannic JM, Blondiaux E, Senat MV, Friszer S, Adamsbaum C, Rousseau J, Hornoy P, Letourneau A, de Laveaucoupet J, Lecarpentier E, Rosenblatt J, Quibel T, Mollot M, Ancel PY, Alison M, Goffinet F. Prognostic value of diffusion-weighted magnetic resonance imaging of brain in fetal growth restriction: results of prospective multicenter study. Ultrasound Obstet Gynecol. 2020 Dec;56(6):893-900. doi: 10.1002/uog.21926. PMID 31765031
- [Background] Thornton JG, Hornbuckle J, Vail A, Spiegelhalter DJ, Levene M; GRIT study group. Infant wellbeing at 2 years of age in the Growth Restriction Intervention Trial (GRIT): multicentred randomised controlled trial. Lancet. 2004 Aug 7-13;364(9433):513-20. doi: 10.1016/S0140-6736(04)16809-8. PMID 15302194
- [Background] Boers KE, Vijgen SM, Bijlenga D, van der Post JA, Bekedam DJ, Kwee A, van der Salm PC, van Pampus MG, Spaanderman ME, de Boer K, Duvekot JJ, Bremer HA, Hasaart TH, Delemarre FM, Bloemenkamp KW, van Meir CA, Willekes C, Wijnen EJ, Rijken M, le Cessie S, Roumen FJ, Thornton JG, van Lith JM, Mol BW, Scherjon SA; DIGITAT study group. Induction versus expectant monitoring for intrauterine growth restriction at term: randomised equivalence trial (DIGITAT). BMJ. 2010 Dec 21;341:c7087. doi: 10.1136/bmj.c7087. PMID 21177352
- [Background] Boyer AC, Goncalves LF, Lee W, Shetty A, Holman A, Yeo L, Romero R. Magnetic resonance diffusion-weighted imaging: reproducibility of regional apparent diffusion coefficients for the normal fetal brain. Ultrasound Obstet Gynecol. 2013 Feb;41(2):190-7. doi: 10.1002/uog.11219. Epub 2013 Jan 3. PMID 22744761